CLINICAL TRIAL: NCT03819543
Title: Transcranial Direct Current Stimulation in SUper REfractory STatus EPilepticus (SURESTEP): Pilot Study of a Novel Therapy in a Common Medical Emergency
Brief Title: SURESTEP: Transcranial Direct Current Stimulation in Super Refractory Status Epilepticus
Acronym: SURESTEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018:133
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2020-11

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Application of transcranial direct current stimulation via scalp electrodes over presumed epileptogenic focus for 20 minutes at 2.0 mA.

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation affects super refractory status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of super refractory status epilepticus
* admitted to the intensive care unit
* identifiable epileptogenic focus on EEG

Exclusion Criteria:

* contraindications to scalp EEG
* lice
* scabies
* other hair/skin infection
* scalp psoriasis
* hypersensitivity
* other severe dermatological condition
* previous adverse reaction to collodion
* vagal nerve stimulator
* implantable cardioverter defibrillator
* cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Ng, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Direct Current Stimulation: Patients receiving transcranial direct current stimulation
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Epileptiform Activity, Per Patient-based
Description: EEG epileptiform activity as defined in units of spikes per second for a given patient. Pre-stim compares spike rates during stimulation to before stimulation. Pre-post compares spike rates after stimulation to before stimulation.
Time Frame: Up to 3 hours per EEG recording
Population: Automated and human counting methods found differing numbers of spikes between patients.
Measure: Median (Inter-Quartile Range); unit: percentage reduction in spikes/sec
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 10
percentage reduction in spikes/sec
  Pre-Stim Change (Automated Counts) | -45.9 [-59 to -11.9]
  Pre-Stim Change (Human Counts): number analyzed (Participants) | 6
  Pre-Stim Change (Human Counts) | -51.6 [-70.2 to -17.9]
  Pre-Post Change (Automated Counts) | -18.3 [-25.4 to -1.4]
  Pre-Post Change (Human Counts): number analyzed (Participants) | 7
  Pre-Post Change (Human Counts) | -25.3 [-42.6 to -15.5]

2. Secondary Outcome: Frequency of Epileptiform Activity, Per-session Based
Description: EEG epileptiform activity as defined in units of spikes per second for a given stimulation session. Pre-stim compares spike rates during stimulation to before stimulation. Pre-post compares spike rates after stimulation to before stimulation.
Time Frame: Up to 3 hours per EEG recording
Population: Automated and human counting methods found differing numbers of spikes between patients.
Measure: Median (Inter-Quartile Range); unit: percentage reduction in spikes/sec
Units Other Than Participants: Sessions
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 10
Number analyzed (Sessions) | 29
percentage reduction in spikes/sec
  Pre-Stim Change (Automated Counts) | -47.2 [-76.8 to -16.7]
  Pre-Stim Change (Human Counts): number analyzed (Participants) | 6
  Pre-Stim Change (Human Counts): number analyzed (Sessions) | 15
  Pre-Stim Change (Human Counts) | -38.5 [-79.7 to -4.7]
  Pre-Post Change (Automated Counts) | -6.8 [-48.7 to 21.5]
  Pre-Post Change (Human Counts): number analyzed (Participants) | 7
  Pre-Post Change (Human Counts): number analyzed (Sessions) | 16
  Pre-Post Change (Human Counts) | -21.8 [-61.4 to 12.7]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 251.1 days
Arm/Group | Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 7/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT03819543/Prot_SAP_000.pdf